CLINICAL TRIAL: NCT00316615
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, Influenza Vaccine, Formulation 2005-2006, When Administered to Non-Elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of a Inactivated Influenza Vaccine When Administered to Non Elderly Adults and Elderly Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71P3S; Eudract number: 2005-000622-23
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Influenza Disease
Keywords: influenza; non elderly adult and elderly; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: influenza vaccine

SUMMARY:
The purpose of this study is to evaluate safety and immunogenicity of a single intramuscular (IM) injection of a Surface Antigen, Inactivated, Influenza Vaccine, Formulation 2005-2006, when Administered to Non-Elderly Adults and Elderly Subjects

ELIGIBILITY:
Inclusion Criteria:

* subjects 18 years of age or older

Exclusion Criteria:

* Any serious disease such as: cancer, autoimmune disease, advanced arteriosclerotic disease or complicated diabetes mellitus, chronic obstructive pulmonary disease (COPD) that requires oxygen therapy, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure
* hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine
* history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
* known or suspected (or high risk of developing) impairment/alteration of immune function

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-06

PRIMARY OUTCOMES:
CHMP criteria for evaluation of flu vaccines e.g Seroprotection, GMR's and Seroconversion rate at day 21 following vaccination

SECONDARY OUTCOMES:
Number and percentage of subjects with at least one local reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one systemic reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one adverse event between Day 0 and the study termination visit (Day 21, window: 20-24).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Drug Information Services, Study Chair — Novartis
Locations (2):
- Italy (2):
  - G. D'Annunzio University, Chieti
  - Office of Hygiene and Public Health, ASL Lanciano, Lanciano